CLINICAL TRIAL: NCT01268540
Title: Comparison of Aspheric Toric & Non-toric Aphakic Intraocular Lenses
Acronym: COAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoya Surgical Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-T240
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Aphakia; Cataract
Keywords: intraocular lens; IOL; cataract; refractive astigmatism; Aspheric; Toric; Hoya; Surgical; Optics; visual acuity
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- NHT15 (Experimental): Aspheric Toric Intraocular Lens Models NHT15
  Interventions: Device: NHT15, NHT30, & NHT53
- FY-60AD (Active Comparator): Aspheric Non-toric Intraocular Lens: Model FY-60AD
  Interventions: Device: FY-60AD
- NHT30 (Experimental): Aspheric Toric Intraocular Lens Model NHT30
  Interventions: Device: NHT15, NHT30, & NHT53
- NHT53 (Experimental): Aspheric Toric Intraocular Lens Models NHT53
  Interventions: Device: NHT15, NHT30, & NHT53

INTERVENTIONS:
Device: FY-60AD — Phacoemulsification cataract extraction followed by implantation of an aspheric non-toric intraocular lens: Model FY-60AD.
  Arms: FY-60AD
Device: NHT15, NHT30, & NHT53 — Phacoemulsification cataract extraction followed by implantation of an aspheric toric intraocular lens: Model NHT15, NHT30, or NHT53.
  Arms: NHT15; NHT30; NHT53

SUMMARY:
The purpose of this multi-center clinical trial is to determine the safety and efficacy of the HSO Toric IOLs for the correction of aphakia and reduction of pre-existing refractive astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with cataract for which phacoemulsification extraction and posterior chamber IOL implantation is indicated
* Have at least one eye that meets the ranges of pre-operative corneal cylinder as specified by this study's guidelines, i.e. corneal cylinder of at least 1.0 D (after accounting for changes in corneal cylinder due to the incision)
* Have potential Best Corrected Visual Acuity of 20/30 or better after implantation of a study lens
* Have clear intraocular media other than cataract
* Have preoperative Best Corrected Visual Acuity equal to 20/40 or worse, with or without a glare source

Exclusion Criteria:

* Have atonic pupils or physiologically small pupils in either eye (unable to dilate to at least 4 mm)
* Have irregular astigmatism in the operative eye, or refractive cylinder resulting only from lenticular astigmatism in the operative eye
* Have corneal pathology potentially affecting corneal topography, or other corneal abnormalities that do or are expected to reduce best corrected visual acuity in the operative eye during the study period
* Have undergone previous refractive corneal surgery in the operative eye
* Have been diagnosed with any degenerative retinal disorders (e.g. soft drusen, macular degeneration or other progressive retinal disorders) in the operative eye that are predicted to cause future visual acuity losses to a level of 20/30 or worse during the postoperative follow-up time requirements of this study

Eligibility criteria not complete. Contact Hoya Surgical Optics, Inc. for more information.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
percent reduction of absolute cylinder | up to 14 months

SECONDARY OUTCOMES:
Lens rotation or misalignment and patient satisfaction | up to 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Kees den Besten, Study Director — Hoya Surgical Optics, Inc.
Locations (6):
- United States (6):
  - Contact Hoya Surgical Optics, Inc. for Trial Locations, Chino Hills, California
  - Shepard Eye Center, Santa Maria, California
  - Mid-Florida Eye Center, Mt. Dora, Florida
  - Grosinger, Spigelman & Grey,, Bloomfield Hills, Michigan
  - Silverstein Eye Conters, Dansas City, Missouri
  - Cleveland Eye Clinic, Brecksville, Ohio